CLINICAL TRIAL: NCT02438696
Title: Relative Bioavailability of Two Newly Developed Tablet Formulations (TF2 and iFF) Compared to BI 1060469 TF1 Formulation, Following Oral Administration (Low and High Dose) in Healthy Female Subjects (an Open-label, Randomised, Single-dose, Three-period, Three-sequence Crossover Study at Two Different Dose Strengths)
Brief Title: Relative Bioavailability of Two Newly Developed Tablet Formulations (TF2 and iFF)Compared to BI 1060469 TF1 Formulation, Following Oral Administration (Low and High Dose)in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1333.4; 2014-005507-24 (EudraCT Number: EudraCT)
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Healthy

ARMS (6):
- 3 BI 1060469 low dose (Experimental): TF2 followed by iFF followed by TF1
  Interventions: Drug: BI 1060469, TF1, Reference; Drug: BI 1060469, TF2, Test; Drug: BI 1060469, iFF, Test
- 1 BI 1060469 high dose (Experimental): TF1 followed by TF2 followed by iFF
  Interventions: Drug: BI 1060469, iFF, Test; Drug: BI 1060469, TF1, Reference; Drug: BI 1060469, TF2, Test
- 2 BI 1060469 high dose (Experimental): iFF followed by TF1 followed by TF2
  Interventions: Drug: BI 1060469, iFF, Test; Drug: BI 1060469, TF2, Test; Drug: BI 1060469, TF1, Reference
- 3 BI 1060469 high dose (Experimental): TF2 followed by iFF followed by TF1
  Interventions: Drug: BI 1060469, TF2, Test; Drug: BI 1060469, iFF, Test; Drug: BI 1060469, TF1, Reference
- 1 BI 1060469 low dose (Experimental): TF1 followed by TF2 followed by iFF
  Interventions: Drug: BI 1060469, iFF, Test; Drug: BI 1060469, TF1, Reference; Drug: BI 1060469, TF2, Test
- 2 BI 1060469 low dose (Experimental): iFF followed by TF1 followed by TF2
  Interventions: Drug: BI 1060469, iFF, Test; Drug: BI 1060469, TF1, Reference; Drug: BI 1060469, TF2, Test

INTERVENTIONS:
Drug: BI 1060469, iFF, Test
  Arms: 2 BI 1060469 high dose
Drug: BI 1060469, iFF, Test
  Arms: 1 BI 1060469 high dose
Drug: BI 1060469, TF1, Reference
  Arms: 3 BI 1060469 low dose
Drug: BI 1060469, TF2, Test
  Arms: 2 BI 1060469 high dose
Drug: BI 1060469, TF2, Test
  Arms: 3 BI 1060469 high dose
Drug: BI 1060469, iFF, Test
  Arms: 2 BI 1060469 low dose
Drug: BI 1060469, TF1, Reference
  Arms: 1 BI 1060469 high dose
Drug: BI 1060469, iFF, Test
  Arms: 3 BI 1060469 high dose
Drug: BI 1060469, iFF, Test
  Arms: 1 BI 1060469 low dose
Drug: BI 1060469, TF1, Reference
  Arms: 2 BI 1060469 low dose
Drug: BI 1060469, TF2, Test
  Arms: 3 BI 1060469 low dose
Drug: BI 1060469, TF1, Reference
  Arms: 2 BI 1060469 high dose
Drug: BI 1060469, TF1, Reference
  Arms: 1 BI 1060469 low dose
Drug: BI 1060469, TF2, Test
  Arms: 1 BI 1060469 high dose
Drug: BI 1060469, TF2, Test
  Arms: 1 BI 1060469 low dose
Drug: BI 1060469, iFF, Test
  Arms: 3 BI 1060469 low dose
Drug: BI 1060469, TF2, Test
  Arms: 2 BI 1060469 low dose
Drug: BI 1060469, TF1, Reference
  Arms: 3 BI 1060469 high dose

SUMMARY:
The primary objective is to investigate the relative bioavailability of two newly developed tablet formulations of BI 1060469 vs BI 1060469 TF1 formulation. The secondary objective is the comparison of several pharmacokinetic parameters between the treatments.

ELIGIBILITY:
Inclusion criteria:

* Healthy female subjects according to the investigator¿s assessment, based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 50 years (incl.)
* BMI of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm at screening
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Intake of drugs with a long half-life (more than 24 h) within 30 days or less than 10 halflives of the respective drug prior to administration of trial medication
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 20 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 470 ms in females) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Positive pregnancy test, pregnancy or plans to become pregnant within 30 days after study completion
* Lactation period

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | up to 72 h
Cmax (maximum measured concentration of the analyte in plasma) | up to 72 h

SECONDARY OUTCOMES:
AUC0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 72 h

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1333.4.1 Boehringer Ingelheim Investigational Site, Biberach, Germany